CLINICAL TRIAL: NCT01716650
Title: A Pilot Study to Evaluate the Contribution of the Saphenous Nerve in Ankle Pain of Patients With Degenerative Joint Disease of the Ankle
Status: Terminated | Type: Observational
Why Stopped: no available participants
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Steven R. Clendenen, Principal Investigator, Mayo Clinic
Other Study IDs: 09-007710
Record Dates: First submitted 2012-10-24; First posted 2012-10-30 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2017-12

CONDITIONS: Degenerative Joint Disease of the Ankle
Keywords: ankle; saphenous nerve block

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Saphenous nerve block: Data collection after saphenous nerve block placement

SUMMARY:
To assess the pain scores before and after saphenous nerve block placement in patients with degenerative joint disease of the ankle

ELIGIBILITY:
Inclusion Criteria:

* Patients evaluated with osteoarthritis who are surgical candidates for ankle fusion or total ankle replacement.
* Registered patients at Mayo Clinic in Florida with scheduled visit to see Dr.Whalen

Exclusion Criteria:

* Patients with lower extremity diabetic neuropathy
* History of prior trauma of ankle with residual nerve injury
* Current medication of pregabalin or gabalin
* Allergy to lidocaine.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with degenerative joint disease of the ankle evaluated in the orthopedic department
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Ankle pain | 30 minutes
  Patient's ankle pain will be assessed prior to and after the nerve block. The study will assess if pain score is lower after the saphenous nerve block

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials